CLINICAL TRIAL: NCT07310602
Title: The Effects of Dim Light (≤80 Lux) Exposure During Labor on Pain, Anxiety, and Labor Progress: A Single-Center Randomized Controlled Trial
Brief Title: Effects of Dim Light During Labor on Pain, Anxiety, and Labor Progress
Acronym: DIM-LIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pınar Erdoğan (Other)
Responsible Party: Sponsor-Investigator, Pınar Erdoğan, MD, Assoc. Prof., Nigde Omer Halisdemir University
Organization: Nigde Omer Halisdemir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/131
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Labor Pain and Anxiety; Labor Progress
Keywords: Dim light; Lighting intensity; Labor room environment; Labor pain; Anxiety during labor; Childbirth; Intrapartum care; Non-pharmacological intervention
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two parallel study groups. To reduce contamination between groups, cluster randomization by delivery room and study week is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dim Light (50-80 Lux) (Experimental): Labor room lighting will be maintained at 50-80 lux using warm white/amber light sources. Illumination will be monitored at regular intervals with a lux meter. Standard intrapartum care will be provided; lighting may be increased immediately if clinically needed.
  Interventions: Other: Dim Light Exposure During Labor
- Routine Lighting (Control) (Active Comparator): Routine labor room lighting will be maintained according to standard clinical practice. Standard intrapartum care will be provided.
  Interventions: Other: Routine Labor Room Lighting

INTERVENTIONS:
Other: Dim Light Exposure During Labor — Adjustment of labor room illumination to a target range of 50-80 lux during active labor, with monitoring using a lux meter; lighting can be increased at any time for clinical reasons.
  Arms: Dim Light (50-80 Lux)
Other: Routine Labor Room Lighting — Standard labor room lighting conditions maintained according to routine clinical practice, without modification of illumination levels.
  Arms: Routine Lighting (Control)

SUMMARY:
The environment of the labor room may influence how women experience childbirth. Light levels, in particular, may affect comfort, stress, and the course of labor. However, there is limited high-quality evidence on whether keeping the labor room lighting dim has measurable benefits for mothers.

This study aims to evaluate the effects of dim light exposure during active labor on pain, anxiety, and labor progress. Pregnant women who are in active labor at term will be randomly assigned to one of two groups. One group will give birth in a room with dim lighting (50-80 lux), while the other group will receive standard room lighting as part of routine care.

Pain and anxiety levels will be measured at specific time points during labor using standard assessment scales. Information about labor duration, use of labor medications, mode of delivery, and newborn outcomes will also be collected.

The dim light intervention does not interfere with routine obstetric care and does not pose additional risk to the mother or baby. If needed for clinical reasons, room lighting can be increased immediately. The results of this study may help determine whether a simple change in the birth environment can improve maternal comfort and labor outcomes.

DETAILED DESCRIPTION:
This study is a single-center, parallel-group randomized controlled trial designed to evaluate the effects of dim light exposure during active labor on maternal pain, anxiety, and labor progress. The trial is conducted in a university hospital labor ward and includes term pregnant women in active labor.

Eligible participants are women aged 18-45 years with a singleton, vertex-presenting pregnancy at ≥37 weeks of gestation who are in active labor. Participants are allocated to one of two study groups according to a predefined randomization scheme. To minimize contamination between groups, cluster randomization by delivery room and week is applied.

In the intervention group, labor room lighting is adjusted to a dim light environment with an illumination level maintained between 50 and 80 lux, using warm white or amber light sources. Light intensity is monitored at regular intervals using a lux meter. In the control group, routine labor room lighting conditions are maintained in accordance with standard clinical practice.

Pain intensity and anxiety levels are assessed at predefined time points during labor using validated measurement tools. Labor progress and obstetric outcomes, including use of labor augmentation, duration of labor stages, mode of delivery, and neonatal outcomes, are recorded from clinical charts.

The primary outcome is derived from changes in pain intensity over time during labor. Secondary outcomes include anxiety levels, labor characteristics, and maternal and neonatal clinical outcomes.

The dim light intervention is non-invasive and does not interfere with routine obstetric care. For clinical or safety reasons, room lighting can be increased immediately at any time at the discretion of the clinical team. All participants receive standard intrapartum care according to institutional protocols.

Study data are collected prospectively and stored in an anonymized format to ensure participant confidentiality. The study is conducted in accordance with ethical principles and has received approval from the relevant institutional ethics committee.

ELIGIBILITY:
Inclusion Criteria:

Pregnant individuals aged 18-45 years

Singleton pregnancy

Vertex (cephalic) presentation

Gestational age ≥37 weeks

Active labor at enrollment (cervical dilation between 4 and 8 cm)

Ability to provide written informed consent

Exclusion Criteria:

Planned or ongoing epidural analgesia

Multiple pregnancy

Severe preeclampsia or other obstetric complications requiring immediate intervention

Known photosensitivity or light-related sensitivity disorders

History of psychiatric disorders that may interfere with anxiety assessment

Any condition deemed by the clinical team to require deviation from the study protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity over time (VAS-AUC, 0-120 minutes) | From baseline to 120 minutes during active labor
  Pain intensity will be assessed using a 0-10 Visual Analog Scale (VAS) at baseline (0 minutes), 60 minutes, and 120 minutes after allocation. The area under the curve (AUC) for VAS from 0 to 120 minutes will be calculated as the primary outcome.

SECONDARY OUTCOMES:
Anxiety level (STAI-S change) | From baseline to 90 minutes during active labor
  State anxiety will be assessed using the State-Trait Anxiety Inventory - State Anxiety Scale (STAI-S) at baseline (prior to intervention/exposure) and at 90 minutes during active labor. The STAI-S consists of 20 items, with total scores ranging from 20 to 80. Higher STAI-S scores indicate greater state anxiety (worse outcome). The primary analysis will use the change score (90-minute STAI-S minus baseline STAI-S); negative values indicate a reduction in anxiety.
Oxytocin use (initiation rate and total dose) | During labor until delivery
  Proportion of participants who receive oxytocin augmentation and the total oxytocin dose administered during labor will be recorded from clinical charts.
Duration of active phase of labor | From enrollment to full dilation
  Time from enrollment during active labor to full cervical dilation will be recorded.
Duration of second stage of labor | From full dilation to delivery
  Time from full cervical dilation to delivery will be recorded.
Mode of delivery | At delivery
  Vaginal delivery (spontaneous/assisted) and cesarean delivery will be recorded.
Estimated blood loss | At delivery / immediate postpartum
  Estimated maternal blood loss at delivery will be recorded from clinical records.
Neonatal outcomes (Apgar scores) | 1 and 5 minutes after birth
  Neonatal well-being will be assessed using the Apgar scoring system at 1 and 5 minutes after birth. The Apgar score ranges from 0 to 10, based on five components (heart rate, respiratory effort, muscle tone, reflex irritability, and skin color). Higher Apgar scores indicate better neonatal condition (better outcome). Apgar scores at 1 and 5 minutes will be recorded and analyzed descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University Hospital, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of intrapartum clinical data and the absence of participant consent for data sharing beyond the objectives of this study. De-identified aggregate results will be reported through publications.

REFERENCES:
- [Background] Zsido AN, Teleki SA, Csokasi K, Rozsa S, Bandi SA. Development of the short version of the spielberger state-trait anxiety inventory. Psychiatry Res. 2020 Sep;291:113223. doi: 10.1016/j.psychres.2020.113223. Epub 2020 Jun 12. PMID 32563747
- [Background] Wronding T, Argyraki A, Petersen JF, Topsoe MF, Petersen PM, Lokkegaard ECL. The aesthetic nature of the birthing room environment may alter the need for obstetrical interventions - an observational retrospective cohort study. Sci Rep. 2019 Jan 22;9(1):303. doi: 10.1038/s41598-018-36416-x. PMID 30670709
- [Background] Balabanoff D. Color, light, and birth space design: An integrative review. Color Res Appl. 2023;48:413-32. doi: 10.1002/COL.22842
- [Background] Kazemi A, Beigi M, Najafabadi HE. Environmental factors influencing women's childbirth experiences in labor-delivery-recovery-postpartum unit: a qualitative cross-sectional study. BMC Pregnancy Childbirth. 2023 Mar 13;23(1):169. doi: 10.1186/s12884-023-05488-7. PMID 36915051
- [Background] Buckley SJ. Executive Summary of Hormonal Physiology of Childbearing: Evidence and Implications for Women, Babies, and Maternity Care. J Perinat Educ. 2015;24(3):145-53. doi: 10.1891/1058-1243.24.3.145. PMID 26834435